CLINICAL TRIAL: NCT00469443
Title: A Randomized Phase III Study of Irinotecan Plus 5-fluorouracil Plus Leucovorin and Bevacizumab (FOLFIRI+Avastin) Versus Irinotecan Plus Capecitabine and Bevacizumab (XELIRI+Avastin) as 1st Line Treatment of Locally Advanced or Metastatic Colorectal Cancer
Brief Title: Randomized Phase III Study of Folfiri+Avastin Versus Xeliri+Avastin as 1st Line Treatment of CRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: J.Sougklakos, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.16
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer; Irinotecan; Capecitabine; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Fluorouracil; Leucovorin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): FOLFIRI/Avastin
  Interventions: Drug: Irinotecan; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Bevacizumab
- 2 (Experimental): XELIRI/Avastin
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 150mg/m2 IV on day 1 every 2 weeks for 10 cycles
  Other Names: CPT-11
  Arms: 1
Drug: 5-Fluorouracil — 5-Fluorouracil 400 mg/m2 infused over 10 min IV and 5-FU 600 mg/m2 infused over 22 hours IV, on Day 1 and 2 (De Grammont regimen), every 2 weeks for 10 cycles
  Other Names: 5-FU
  Arms: 1
Drug: Leucovorin — Leucovorin 200 mg/m2 infused over 2 hours IV, on day 1 and 2 every 2 weeks for 10 cycles
  Other Names: LV
  Arms: 1
Drug: Capecitabine — Capecitabine 2000mg/m2 p.o. daily, for days 1-14, every 3 weeks for 6 cycles
  Other Names: Xeloda
  Arms: 2
Drug: Bevacizumab — Bevacizumab 5mg/kg IV on day 1 every 2 weeks for 10 cycles
  Other Names: Avastin
  Arms: 1
Drug: Bevacizumab — Bevacizumab 7,5mg/kg IV on day 1 every 3 weeks for 6 cycles
  Other Names: Avastin
  Arms: 2
Drug: Irinotecan — Irinotecan 250mg/m2 IV on day 1 every 3 weeks for 6 cycles
  Other Names: CPT-11
  Arms: 2

SUMMARY:
This phase III study will compare two combinations of irinotecan, Folfiri versus Xeliri, with the addition of Avastin as 1st line treatment of colorectal cancer.

DETAILED DESCRIPTION:
There is no data of comparison for Folfiri and Xeliri regimens. The reported data demonstrated that the addition of Avastin in the combination of irinotecan/bolus 5-FU/LV has significant improvement of overall survival. Further analysis of these results showed that patients receiving irinotecan in combination with Avastin, as 1st line treatment and oxaliplatin with Avastin, as second line treatment, have median overall survival 25, 1 months, which is the longest survival that has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal cancer
* Measurable or evaluable disease
* ECOG performance status ≤ 2
* Age 18 - 72 years
* Adequate liver (Bilirubin ≤ 1.5 UNL, SGOT/SGPT ≤ 4 UNL, ALP ≤ 2.5 UNL), renal (Creatinine ≤ 1.5 UNL) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥ 100,000/mm3) function
* Patients with history of hemoptysis or with increased risk of thromboembolic events should be observed carefully due to administration of Avastin
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* Previous 1st line chemotherapy
* Adjuvant chemotherapy with Irinotecan regimen with relapse < 6 months after the completion
* Active infection
* History of serious cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow
* Patients with unstable CNS metastases
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women
* Patients > 65 years with history of arterial thromboembolic, myocardial infarction, unstable angina and pulmonary embolism

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Time To Progression | 1 year

SECONDARY OUTCOMES:
Objective Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Overall Survival | Probability of 1-year survival (%)
Toxicity profile | Toxicity assessment on each chemotherapy cycle
Quality of life | Assessment every two cycles
Symptoms improvement | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — johnsougl@gmail.com
Locations (8):
- Greece (8):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Souglakos J, Ziras N, Kakolyris S, Boukovinas I, Kentepozidis N, Makrantonakis P, Xynogalos S, Christophyllakis Ch, Kouroussis Ch, Vamvakas L, Georgoulias V, Polyzos A. Randomised phase-II trial of CAPIRI (capecitabine, irinotecan) plus bevacizumab vs FOLFIRI (folinic acid, 5-fluorouracil, irinotecan) plus bevacizumab as first-line treatment of patients with unresectable/metastatic colorectal cancer (mCRC). Br J Cancer. 2012 Jan 31;106(3):453-9. doi: 10.1038/bjc.2011.594. Epub 2012 Jan 12. PMID 22240792